CLINICAL TRIAL: NCT04667013
Title: A Bridged Phase 1, Randomized, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of TBN in Healthy Subjects
Brief Title: A Multiple Dose Study to Investigate Safety, Tolerability and Pharmacokinetics of TBN
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Magpie Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 192008
Record Dates: First submitted 2020-12-01; First posted 2020-12-14 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Phase 1; Amyotrophic lateral sclerosis; TBN
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — tetramethylpyrazine nitrone; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 2 x 300 mg TBN tablets for a total dose of 600 mg or 2 matching placebo tablets (given approximately every 12 hours) for 6.5 consecutive days, until the morning dose of Day 7.
  Interventions: Drug: Tetramethylpyrazine nitrone (TBN) tablet / Placebo
- Cohort 2 (Experimental): 4 x 300 mg TBN tablets for a total dose of 1200 mg or 4 matching placebo tablets (given approximately every 12 hours) for 6.5 consecutive days, until the morning dose of Day 7.
  Interventions: Drug: Tetramethylpyrazine nitrone (TBN) tablet / Placebo

INTERVENTIONS:
Drug: Tetramethylpyrazine nitrone (TBN) tablet / Placebo — Subjects will be administered multiple oral doses of TBN or matching placebo tablets twice a day for 6 consecutive days and a last dose in the morning of Day 7.
  Other Names: TBN tablet / Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics (i.e. how study drug is taken up by the body) of TBN in healthy participants.

DETAILED DESCRIPTION:
The trial is a single center, placebo-controlled, double-blind, multiple-dose study in 2 ascending dose cohorts of healthy subjects. The primary purpose of this study is to investigate the safety, tolerability and pharmacokinetic property of the multiple doses of TBN administered for 6.5 consecutive days in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-childbearing potential female, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥ 18 and ≤ 50 years of age, with BMI > 18.0 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Healthy as defined by:

   1. The absence of clinically significant illness and surgery within 4 weeks prior to the first dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Investigator.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Non-childbearing potential female is defined as:

   1. Post-menopausal female (absence of menses for 12 months prior to the first study drug administration, bilateral oophorectomy or hysterectomy with bilateral oophorectomy at least 6 months prior to the first study drug administration);

      or
   2. Surgically sterile female (hysterectomy or tubal ligation at least 6 months prior to drug administration).
4. Male subjects who have not been vasectomized for at least 6 months prior, and who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration:

   1. Simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks prior or intra-uterine contraceptive device placed since at least 4 weeks prior;
   2. Simultaneous use of a male condom and, for the female partner, a diaphragm or cervical cap with intravaginally applied spermicide.
5. Male subjects (including men who have had a vasectomy) with a pregnant partner must agree to use a condom from the first study drug administration until at least 90 days after the last study drug administration.
6. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
7. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen, alcohol breath test, or urine cotinine test at screening.
3. History of allergic reactions to TBN or other related drugs, or to any excipient in the formulation.
4. Positive pregnancy test at screening.
5. Clinically significant ECG abnormalities or vital sign abnormalities, systolic BP lower than 90 or over 140 mmHg, diastolic BP lower than 50 or over 90 mmHg, or heart rate (HR) less than 50 or over 100 bpm; orthostatic BP: decrease in systolic BP of 20 mmHg or higher, decrease in diastolic BP of 10 mmHg or higher, or increase in HR of 30 bpm or higher within 2 to 3 minutes after passing from a supine to a standing position at screening.
6. History of significant alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit (more than 14 units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
7. History of significant drug abuse within 1 year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine (PCP), crack, opioid derivatives including heroin, and amphetamine derivatives) within 1 year prior to screening.
8. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
9. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the pharmacokinetics (PK) profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

   1. Prescription medications within 14 days prior to the first dosing;
   2. Over-the-counter products and natural health products (including herbal remedies, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
   3. Depot injection or implant of any drug within 3 months prior to the first dosing;
   4. Any drugs known to induce or inhibit hepatic drug metabolism (including St. John's wort) within 30 days prior to the first dosing.
10. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
11. Any reason which, in the opinion of the Investigator, would prevent the subject from participating in the study.
12. Breast-feeding subject.
13. Any history of thyroid/gland abnormalities.
14. Any history of suicidal ideation or suicidal behavior (within 2 years prior to screening), as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) (baseline version).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | 14 days
  The number and severity of AEs will be graded according to criteria from the NCI-CTCAE (i.e., seriousness, severity, relationship to the study medication, outcome, duration, and management).
Assessment of physical examination. | 14 days
  Physical examination will be assessed on Day-1, Day4, and check-out (Day8), follow-up visit (Day14±2).
Assessment of vital signs. | 14 days
  Vital signs, including orthostatic blood pressure and heart rate, respiratory rate and oral temperature, will be evaluated from Day-1 to check-out (Day8), and at follow-up visit (Day14±2).
Assessment of 12 lead-ECG. | 14 days
  12 lead-ECG will be assessed on Day-1, Day4, Day 7 and at check-out (Day8), follow-up visit (Day14±2).
Assessment of urine pregnancy. | 14 days
  Urine pregnancy test will be assessed on Day-1 and at follow-up visit (Day14±2).
Assessment of Clinical Laboratory Tests. | 14 days
  Clinical laboratory tests includes hematology, clinical chemistry, coagulation (prothrombin time and partial thromboplastin time), endocrinology (T3, T4, and thyroid stimulating hormone) and urinalysis, will be assessed on Day-1, Day2, Day4, Day6 and at check-out (Day8), follow-up visit (Day14±2).

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of TBN and its metabolite. | 0 to 12 hours after on the morning dosing of the first day
  Plasma concentrations of TBN and its metabolite [Time point: pre-dose, 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 (prior to the second dose)], and derived pharmacokinetic parameters Cmax.
Time of occurrence of Cmax (Tmax) of TBN and its metabolite. | 0 to 12 hours after on the morning dosing of the first day
  Plasma concentrations of TBN and its metabolite [Time point: pre-dose, 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 (prior to the second dose)], and derived pharmacokinetic parameters Tmax.
Area under the concentration-time curve from time zero to time 12 hours (AUC0-12) of TBN and its metabolite. | 0 to 12 hours after on the morning dosing of the first day
  Plasma concentrations of TBN and its metabolite [Time point: pre-dose, 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12 (prior to the second dose)], and derived pharmacokinetic parameters AUC0-12.
Lowest concentration before the next dose is administered (Ctrough) of TBN and its metabolite. | From Day2 to Day6
  Time point: pre-morning dose of Day2, Day3, Day4, Day5 and Day6.
Area under the concentration-time curve for one dosing interval (12 hours) at steady-state (AUC0-tau) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters AUC0-tau.
Average drug concentration calculated at AUC0-tau/tau (Caverage) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: Time frame: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters Caverage.
Minimum observed concentration at steady-state (Cmin_ss) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: Time frame: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters Cmin_ss.
Area under the concentration-time curve from time zero to the 24 hours concentration (AUC0-24) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: Time frame: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters AUC0-24.
Maximum observed concentration at steady-state (Cmax_ss) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: Time frame: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters Cmax_ss.
Time of observed Cmax_ss (Tmax_ss) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: Time frame: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters Tmax_ss.
Area under the concentration-time curve from time zero to infinity (AUC0-inf) of TBN and its metabolite. | 0-24 hours after the last dose at Day7
  Plasma concentrations of TBN and its metabolite [Time point: Time frame: pre-dose, and 1, 1.5, 1.75, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 10, 12, 14, and 24 hours after the last dose at Day7], and derived pharmacokinetic parameters AUC0-inf.

CONTACTS AND LOCATIONS:
Overall Officials: David Wyatt, VP, Principal Investigator — Syneos Health Inc.

IPD SHARING:
Plan to Share IPD: No